CLINICAL TRIAL: NCT02077231
Title: Study of Vitamin A and Carbomer in Comforting the Ocular Surface Irritations of Glaucoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaodong Zhou (Other)
Responsible Party: Sponsor-Investigator, Xiaodong Zhou, Professor of Ophthalmology, Shanghai Jinshan Hospital
Organization: Shanghai Jinshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GlaucomaVitaminA
Record Dates: First submitted 2014-02-23; First posted 2014-03-04 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Primary Open-angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Vitamin A

ARMS (2):
- vitamin A palmitate eye gel (Experimental): 0.1% vitamin A palmitate; Sinqi, Shenyang, China
  Interventions: Drug: Vitamin A
- carbomer eye gel (Experimental): 0.2% Carbomer 940; Bausch & Lomb, Aschheim, Germany
  Interventions: Drug: carbomer eye gel

INTERVENTIONS:
Drug: Vitamin A — use one drop in the eye
  Other Names: vitamin A palmitate eye gel
  Arms: vitamin A palmitate eye gel
Drug: carbomer eye gel — use one drop in the eye
  Other Names: Carbomer Eye Drops
  Arms: carbomer eye gel

SUMMARY:
Most of the patients under long application of anti-glaucoma eyedrops endure severe ocular surface irritation, which interrupt their quality of life a lot. Lots of studies aimed to search for new drugs for therapy. The investigators hypothesized that the artificial tears containing vitamin A or carbomer may be a great substitute. Both of the two drugs were in common use and had already been tested in animals.

ELIGIBILITY:
Inclusion Criteria:

- diagnosed primary open-angle glaucoma or normal tension glaucoma patients with prostaglandin analogs treatment for more than one year.

Exclusion Criteria:

1. any systemic diseases which may cause ocular damage;
2. previous ocular trauma or surgery;
3. contact lens wear history in previous 6 months;
4. application of any artificial tears 3 months ago;
5. allergic to any of the drugs we used during examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-09; Primary Completion 2013-02 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
change of the density of conjunctival goblet cells | change from Baseline in goblet cell density at 6 months

SECONDARY OUTCOMES:
tear film parameters changes in patients | change from baseline in TBUT and Schirmer test at 6 months
changes of ocular irritation in patients | change from baseline in OSDI scores at 6 months